CLINICAL TRIAL: NCT02061865
Title: Phase 1 Safety Study With Intravitreal (IVT) REGN2176-3 in Patients Aged 50 Years and Older With Wet AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2176-3-AMD-1303
Record Dates: First submitted 2014-01-28; First posted 2014-02-13 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Neovascular Wet Age-related Macular Degeneration (AMD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohorts 1 - 4 (Experimental): Participants in cohort 1 will receive REGN2176-3 dosing regimen 1. Participants in cohort 2 will receive REGN2176-3 dosing regimen 2. Participants in cohort 3 will receive REGN2176-3 dosing regimen 3. Participants in cohort 4 will receive REGN2176-3 dosing regimen 4.
  Interventions: Drug: REGN2176-3

INTERVENTIONS:
Drug: REGN2176-3

SUMMARY:
The primary objective of the study is to investigate the safety of intravitreal (IVT) REGN2176-3 in patients with neovascular wet age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

Key Criteria:

Men or women greater than or equal to 50 years of age who provide informed consent and have active subfoveal choroidal neovascularization (CNV) secondary to wet AMD.

Exclusion Criteria:

1. Any prior treatment with an inhibitor of PDGF (platelet-derived growth factor) or PDGFR (platelet-derived growth factor receptor)
2. Active neovascular AMD in the fellow eye requiring treatment
3. Scar, fibrosis, or atrophy in the study eye involving the center of the fovea
4. Presence of retinal pigment epithelial tears or rips involving the macula in the study eye
5. Prior vitrectomy in the study eye
6. Any history of macular hole of stage 2 and above in the study eye
7. Any intraocular or periocular surgery within 3 months of day 1 in the study eye, except lid surgery
8. History of corneal transplant in the study eye
9. Positive serum human chorionic gonadotropin (hCG)/ urine pregnancy test at the screening or baseline visit

The information listed above is not intended to contain all considerations relevant to a patient's potential participation in this clinical trial and not all inclusion/ exclusion criteria are listed.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety | day 1 through week 24
  The primary endpoint in the study is the incidence of treatment emergent adverse events (TEAEs) from day 1 through week 24 in patients treated with IVT REGN2176-3.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (4):
- United States (4):
  - Beverly Hills, California
  - Colorado Springs, Colorado
  - Boston, Massachusetts
  - Houston, Texas